CLINICAL TRIAL: NCT00005552
Title: Isocyanate Dermal Exposures in Autobody Shops
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5096; R01HL062932 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To characterize the skin route of exposure to the allergen hexamethylene diisocyanate (HDI) in the auto body industry.

DETAILED DESCRIPTION:
BACKGROUND:

Isocyanates account for the highest number of reported cases of occupational asthma in the United States and developed countries. Prevention, however is limited by inadequate knowledge of isocyanate routes of exposure, exposure patterns, mechanisms of sensitization and other causal factors. The Survey of Painters and Repairers of Auto Bodies by Yale (SPRAY), a five-year cross-sectional epidemiologic survey of painters and repairers of autobodies at Yale was therefore initiated to address these questions. At the outset of Spray, it was not known how frequent skin contact among the painters might be. Moreover, there is new and exciting data from animal studies demonstrating that dermal rather than respiratory contact may be crucial to immune sensitization leading to asthma. Little is known, so far, about dermal exposure in autobody shops and its modifiers, especially the effectiveness of personal protective equipment (PPE) in preventing workers from skin contamination by isocyanates.

DESIGN NARRATIVE:

The study was ancillary to the SPRAY study and was integrated into it. The overall design was a cross-sectional investigation of 20 shops with 120 workers. This would allow a better understanding of the complex basis for asthma risk in these workers, and better recommendations to autobody shops and workers on protective measures for isocyanate dermal exposures.

Specific aims included: 1) Qualitatively and quantitatively assessing surface and skin contamination of HDI; 2) Identifying modifiers that affected surface and skin contamination, and specifically evaluating the effectiveness of personal protective equipment in protecting the skin from isocyanate contamination; 3) Exploring the relationships of dermal exposure with airborne exposure, biomarkers of systemic absorption and skin sensitization, and asthma-developing risk.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cullen — Yale University

REFERENCES:
- [Background] Liu Y, Sparer J, Woskie SR, Cullen MR, Chung JS, Holm CT, Redlich CA. Qualitative assessment of isocyanate skin exposure in auto body shops: a pilot study. Am J Ind Med. 2000 Mar;37(3):265-74. doi: 10.1002/(sici)1097-0274(200003)37:33.0.co;2-o. PMID 10642416